CLINICAL TRIAL: NCT05753475
Title: DOES HEMODYNAMIC REGULATION AFFECTS GRAFT FUNCTIONS DURING RENAL TRANSPLANT?
Brief Title: HOW DOES HEMODYNAMIC REGULATION AFFECTS GRAFT FUNCTIONS DURING RENAL TRANSPLANTATION?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Principal investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-23-3249
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Renal Transplant Failure and Rejection; Hypotension
MeSH Terms: conditions — Rejection, Psychology; Hypotension | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypotension
  Interventions: Other: renal transplantation
- normotension
  Interventions: Other: renal transplantation

INTERVENTIONS:
Other: renal transplantation — patients undergoing renal transplantation

SUMMARY:
The aim of the researchers was to evaluate the adequacy of graft function in the postoperative period of patients who underwent renal transplantation and encountered hypotension in the intraoperative period.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing renal transplantation

Exclusion Criteria:

* patient refusal

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing renal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | baseline
Mean Arterial Pressure | baseline
Systolic Blood Pressure | during the surgery
Mean Arterial Pressure | during the surgery
graft function | immediately after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided